CLINICAL TRIAL: NCT02972164
Title: Adapted Cognitive Behavioural Approach to Addressing Overweight and Obesity Among Qatari Youth
Brief Title: Adapted Cognitive Behavioral Approach to Addressing Overweight and Obesity Among Qatari Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qatar University (Other)
Collaborators: Imperial College London (Other); Hamad Medical Corporation (Industry); Supreme Council Of Health, Qatar (Other Government); Aspetar (Other); Leeds Beckett University (Other)
Responsible Party: Principal Investigator, Prof. Mohamed Ahmedna, Professor, Qatar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X - 036 - 3 - 013
Record Dates: First submitted 2016-11-14; First posted 2016-11-23 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Obesity
Keywords: Childhood obesity; Lifestyle; Prevention; Intervention; Behavioural psychology
MeSH Terms: conditions — Obesity; Pediatric Obesity | interventions — Weight Reduction Programs

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Each year, 100 school children age 9-12 who meet inclusion criteria are selected from 5 randomly chosen schools to participate in the control group. Control children are assessed for the same measures as the intervention group at the beginning and end of the intervention but receive none of the intervention modules.
- Weight loss program for school children (Experimental): Each year, 100 school children age 9-12 who meet inclusion criteria are selected from 5 randomly chosen schools to participate in the intervention group. The intervention children take part in the integrated approach for weight management consisting of (1) intensive weight loss camp (2) twelve weeks of after school clubs for consolidation purposes, and (3) social media and wearable sensors for support and monitoring.
  Interventions: Behavioral: Weight loss program for school children

INTERVENTIONS:
Behavioral: Weight loss program for school children — The intervention involves developing social and emotional competences, promotion of healthy lifestyle, use of activity monitoring devices to promote increased activity and enlisting family to maintain weight loss in the long term.
  The intervention group receives all program components: 1. Parent information sessions and orientation, 2. Two week intensive weight loss and lifestyle education camp, 3. after school clubs for consolidation (including physical activity and lifestyle education), and 4. wearable sensors and social media modules with parental involvement. Assessed outcomes include pre- and post-measurement at each phase included: weight, height, BMI, waist circumference, blood pressure, physical activity, dietary intakes, self-esteem, and subjective well-being.
  Other Names: Cognitive Behavioural and lifestyle
  Arms: Weight loss program for school children

SUMMARY:
Levels of overweight and obesity have reached alarming proportions in Qatar and other Gulf nations. In Qatar, the need to establish national strategies for the prevention and treatment of obesity has been recognized in the new Qatar National Health Strategy 2011-2016, which stresses the need for prevention. In fact, the Qatar National Nutrition and Physical Activity Action Plan 2011-2016 calls for nutrition and physical activity interventions for the prevention of obesity and related chronic diseases such as diabetes. The treatment and prevention of childhood obesity is largely through lifestyle changes- encouraging health eating and physical activity and discouraging sedentary behavior. However, changing such behaviors is complex and requires a combination of integrated approaches to tackle such a multifaceted problem. Herein, the investigators set out to implement and evaluate a novel weight management program for Qatari school children at the vulnerable age of 9-12 years. The project incorporates a cognitive-behavioral approach that involves developing social and emotional competences, promotion healthy dietary habits, development of physical literacy, and use of activity monitoring devices to promote increased activity while enlisting family involvement in an attempt to maintain weight loss in the long term. This project seeks to also take things further by integrating a range of interventions that use cutting edge insights from the behavioral sciences through the use of MINDSPACE approach (MINDSPACE: Messenger, Incentive, Norms, Default, Salience, Priming, Affect, Commitment, Ego) in conjunction with technology tools for monitoring activity and providing ongoing support through the use of social media. The intervention involves a multi-cohort intervention involving 500 Qatari children over 5 years to be conducted in three phases (1) intensive weight loss camps, (2) after-school clubs as supplement/consolidation, and (3) maintenance through web and social/family support.

DETAILED DESCRIPTION:
The specific objectives of the project are to:

1. Adapt and pilot a school-based intervention that combines behavioral and cognitive approaches to promote healthy lifestyle among 9-12 year old children in select Qatari schools in the first year;
2. Integrate behavioral economics and cognitive behavioral therapy (MINDSPACE) in a multi-cohort prevention/intervention study targeting at risk Qatari school children at the vulnerable age range of 9-12;
3. Select and use technological tools for enhanced outcomes and adoption of the intervention nationally;
4. Package study findings into a lifestyle change intervention for national implementation in collaboration with Hamad Medical Corporation and the Supreme Education Council.

Data from this project could provide the basis for a national program to stem the rise of obesity in Qatar through lifestyle changes and reduce related health conditions.

ELIGIBILITY:
Inclusion Criteria:

* School children within age range of 9-12 yrs, at or above 95th percentile of BMI by age using International Obesity TaskForce (IOTF) cut off, and parental consent.

Exclusion Criteria:

* Psychiatric or neurological disorders, learning disability, dyslexia, current or past drug abuse, head injury and psychotropic medication.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 799 (Actual)
Dates: Start 2013-08; Primary Completion 2017-09 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Weight loss | 26 weeks
  Weight loss will be assessed by measurement of Body Mass Index (BMI, expressed in kg/m^2, weight in kilograms, height in meters) at baseline (Day 1 of week 1), post camp (week 3), post clubs (week 14), and post maintenance/end of intervention (week 26). Change in BMI Standard Deviation Scores (SDS) between baseline and week 26 will be used as indicator of effectiveness of intervention compared to BMI-SDS for the control group. One year follow up of change in BMI-SDS for intervention and control groups will gauge the long term benefits of the intervention. A multilevel mixed effects model will be used to assess both individual- (fixed effects) and school-level (random) effects, including covariates, such as demographic factors of the children and time (cohort). BMI SDS will be evaluated to determine mean differences and the proportions of children with significant changes in BMI-SDS throughout the course of the study. Subgroup analyses will be conducted by gender and age.

SECONDARY OUTCOMES:
Adoption of healthier dietary habits | 26 weeks
  This will be measured by administration of a dietary intakes/habits questionnaire using the Children's Dietary Questionnaire at baseline and end of intervention (week 26). The same questionnaire will be administered to the control group for inferential purposes.
Increased physical activity patterns | 26 weeks
  Increased physical activity patterns will be assessed through administration of Physical Activity Questionnaire (PAQ-C) at baseline and end of intervention (week 26). The same questionnaire will be administered to the control group for inferential purposes.
Improvement in self-esteem | 26 weeks
  Self-esteem will be assessed using Rosemberg self-esteem scale at baseline and end of intervention (week 26). The same questionnaire will be administered to the control group for inferential purposes.
Change in impulsivity | 26 weeks
  Changes in impulsivity and subjective wellbeing will be measured using CANTAB Stop Signal Task system at baseline and end of intervention (week 26). The same questionnaire will be administered to the control group for inferential purposes.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ahmedna, PhD, Principal Investigator — Qatar University
Locations (1):
- Qatar University, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vlaev I, Taylor MJ, Taylor D, Gately P, Gunn LH, Abeles A, Kerkadi A, Lothian J, Jreige SK, Alsaadi A, Al-Kuwari MG, Ghuloum S, Al-Kuwari H, Darzi A, Ahmedna M. Testing a multicomponent lifestyle intervention for combatting childhood obesity. BMC Public Health. 2021 Apr 29;21(1):824. doi: 10.1186/s12889-021-10838-1. PMID 33926412
- [Derived] Fernandez-Luque L, Singh M, Ofli F, Mejova YA, Weber I, Aupetit M, Jreige SK, Elmagarmid A, Srivastava J, Ahmedna M. Implementing 360 degrees Quantified Self for childhood obesity: feasibility study and experiences from a weight loss camp in Qatar. BMC Med Inform Decis Mak. 2017 Apr 13;17(1):37. doi: 10.1186/s12911-017-0432-6. PMID 28403865